CLINICAL TRIAL: NCT04708886
Title: Effects of Romosozumab on Bone Health in Women With Spinal Cord Injury and Osteoporosis
Brief Title: Romosozumab in Women With Chronic SCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Thomas J. Schnitzer, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00212405; 20197268 (Other: Amgen Inc.)
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Osteoporosis; Bone Loss; Osteopenia, Osteoporosis; Spinal Cord Injuries; Chronic Spinal Paralysis
Keywords: Spinal Cord Injury; Osteoporosis; Romosozumab (Evenity); Alendronate (Fosamax); Bone Diseases; Metabolic Bone Diseases; Anabolic Treatment; Bisphosphonate; Bone Density; Spinal Cord Diseases; Romosozumab; Alendronate; Physiological Effects of Drugs
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Spinal Cord Injuries; Bone Diseases; Spinal Cord Diseases | interventions — romosozumab; Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Females with Chronic SCI (Experimental): 12-month treatment with monthly subcutaneous romosozumab injections (210 mg), followed by 12-month treatment with weekly oral alendronate tablets (70 mg)
  Interventions: Drug: Romosozumab; Drug: Alendronate

INTERVENTIONS:
Drug: Romosozumab — Year 1 study drug
  Other Names: Evenity
Drug: Alendronate — Year 2 study drug
  Other Names: Fosamax

SUMMARY:
This two-year open-label pilot clinical trial will evaluate the efficacy and safety of romosozumab to treat bone loss in females with chronic spinal cord injury (SCI) and osteoporosis (OP). Participants will receive monthly injections of romosozumab during the first 12 months of the study. During the second year, participants will take oral alendronate tablets on a weekly basis.

DETAILED DESCRIPTION:
This is a single-site, singe-arm, open-label pilot study to evaluate safety and efficacy of a sequential drug treatment (12 months of romosozumab injections followed by 12 months with alendronate tablets) to treat bone loss in women with chronic SCI and OP.

During the first year, participants will receive monthly subcutaneous injections of romosozumab 210 mg. This drug works by increasing bone formation and is FDA-approved for treating OP in post-menopausal women at high risk of fracture or those who did not benefit from using other available OP treatments. During the second year, participants will take weekly oral alendronate 70 mg. Alendronate is FDA-approved for the treatment of osteopenia and the treatment of OP in post-menopausal women and men as well as for the prevention and treatment of glucocorticoid-induced OP. In this study, it will be used to help maintain any increases in bone mass gained from the year of treatment with romosozumab.

Twelve participants will receive the study drug treatment, take daily supplements (calcium and vitamin D), and return to the research site for study visits over the course of two years. Computerized tomography (CT) imaging, dual-energy X-ray absorptiometry (DXA) imaging, and serum bone markers will be collected at various time points.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Female sex
* SCI 6 or more months prior to enrollment
* Non-ambulatory status (Walking Index for Spinal Cord Injury II score of 3 or less)
* Osteoporosis by DXA defined as a t-score of -2.5 at any skeletal site (lumbar spine, total hip, or femoral neck) or a t-score of -2.0 plus a history of a fragility fracture
* Good general health, as determined by the study investigator
* Able to understand and agree to informed consent in English
* Able and willing to complete all the study visits
* Females of childbearing potential must be willing and able to use an effective method of contraception or practice abstinence throughout the course of the study and up to 90 days after the last use of study drug.
* Vitamin D 25-hydroxy levels ≥ 20 ng/ml (subjects may be repleted and retested prior to baseline)
* Normal serum calcium levels (based on current local laboratory normal range)
* No known endocrinopathies (diabetes type 1 or 2, treated thyroid conditions can be included)
* Normal serum thyroid stimulating hormone and/or T4 levels (based on current local laboratory normal ranges)
* Able to take oral medication sitting upright for at least 30 minutes

Exclusion criteria:

* Have Paget's disease of the bone
* Have abnormal laboratory values that in the judgement of the investigator would put the participant at increased risk of treatment
* Any active gastrointestinal condition that results in malabsorption
* Abnormalities of the esophagus which delay emptying such as stricture or achalasia
* Known hypersensitivity to romosozumab or alendronate
* Increased risk of aspiration
* Osteonecrosis of the jaw (ONJ) or risk factor for ONJ, such as invasive dental procedures (e.g., tooth extraction, dental implants, oral surgery in the past 6 months), poor oral hygiene, periodontal and/or pre-existing dental disease, or planned invasive dental procedure over the next two years
* Heterotopic ossification of the knee region that interferes with CT analysis
* History of bone metastasis and skeletal malignancies
* History of alcoholism or drug abuse within the 2 years prior to study screening, which in the opinion of the investigator may affect subject's health and/or study commitment
* Other medical conditions that in the opinion of the investigator would preclude the subject from completing the study
* Currently being prescribed anticonvulsants at a dose or frequency that is determined to interfere with bone metabolism as determined by the investigator
* Currently being prescribed glucocorticoids, other than inhaled glucocorticoids
* Current or use during past 5 years of any bone-active agents, including any FDA approved treatment (e.g., teriparatide, abaloparatide, denosumab, any bisphosphonate (oral or IV), raloxifene, bazedoxifene, hormone therapy (estrogen and estrogen/progestin) and calcitonin) as well as any strontium-containing compounds.
* Pregnant, planning to become pregnant, or lactating
* Any history of stroke or cardiovascular disease other than controlled hypertension
* Renal insufficiency (calculated creatinine clearance less than 35 ml/min)
* Any other neurological impairment that may impair ambulation or muscle function

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Schnitzer, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cosman F, Crittenden DB, Adachi JD, Binkley N, Czerwinski E, Ferrari S, Hofbauer LC, Lau E, Lewiecki EM, Miyauchi A, Zerbini CA, Milmont CE, Chen L, Maddox J, Meisner PD, Libanati C, Grauer A. Romosozumab Treatment in Postmenopausal Women with Osteoporosis. N Engl J Med. 2016 Oct 20;375(16):1532-1543. doi: 10.1056/NEJMoa1607948. Epub 2016 Sep 18. PMID 27641143
- [Background] Saag KG, Petersen J, Brandi ML, Karaplis AC, Lorentzon M, Thomas T, Maddox J, Fan M, Meisner PD, Grauer A. Romosozumab or Alendronate for Fracture Prevention in Women with Osteoporosis. N Engl J Med. 2017 Oct 12;377(15):1417-1427. doi: 10.1056/NEJMoa1708322. Epub 2017 Sep 11. PMID 28892457
- [Background] Keaveny TM, Crittenden DB, Bolognese MA, Genant HK, Engelke K, Oliveri B, Brown JP, Langdahl BL, Yan C, Grauer A, Libanati C. Greater Gains in Spine and Hip Strength for Romosozumab Compared With Teriparatide in Postmenopausal Women With Low Bone Mass. J Bone Miner Res. 2017 Sep;32(9):1956-1962. doi: 10.1002/jbmr.3176. Epub 2017 Jun 26. PMID 28543940

RESULTS

PARTICIPANT FLOW:
Groups:
- Females With Chronic SCI: 12-month treatment with monthly subcutaneous romosozumab injections (210 mg), followed by 12-month treatment with weekly oral alendronate tablets (70 mg).
  Romosozumab was the investigational drug for Year 1; alendronate was administered as standard-of-care in Year 2.
Period: Year 1: Romosozumab
Arm/Group | Females With Chronic SCI
Started | 12
Completed | 12
Not Completed | 0
Period: Year 2: Alendronate
Arm/Group | Females With Chronic SCI
Started | 12
Completed | 10
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Open-label Romosozumab: Participants received monthly subcutaneous injections of romosozumab (210 mg) for 12 months.
Arm/Group | Open-label Romosozumab
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Integral vBMC at the Knee (Distal Femur)
Description: Change from baseline to the Month 12 visit in volumetric bone mineral content (vBMC) obtained via CT (three-dimensional) imaging of the knee.
Time Frame: Baseline - 12 months
Population: Females with Chronic SCI
Measure: Median (Inter-Quartile Range); unit: g
Groups:
- Females With Chronic SCI: Participants received monthly subcutaneous injections of romosozumab (210 mg) for 12 months, followed by weekly oral alendronate (70 mg) for an additional 12 months.
  Romosozumab was the investigational drug for Year 1; alendronate was administered as standard-of-care in Year 2.
Arm/Group | Females With Chronic SCI
Number analyzed (Participants) | 12
g | -0.78 [-1.93 to -0.60]

2. Secondary Outcome: Change in BMD at the Total Hip and Femoral Neck
Description: Change from baseline to the Month 12 visit in bone mineral density (BMD) obtained via DXA (two-dimensional) imaging of the total hip.
Time Frame: Baseline - 12 months
Population: Females with Chronic SCI
Measure: Median (Inter-Quartile Range); unit: g/cm^2
Arm/Group | Females With Chronic SCI
Number analyzed (Participants) | 12
g/cm^2
  Total Hip | 0.023 [0.016 to 0.033]
  Femoral Neck | 0.033 [0.008 to 0.049]

3. Secondary Outcome: Change in vBMC at the Hip
Description: Change from baseline to the Month 12 visit in volumetric bone mineral content (vBMC) obtained via CT imaging of the hip.
Time Frame: Baseline - 12 months
Population: Females with Chronic SCI
Measure: Median (Inter-Quartile Range); unit: g
Arm/Group | Females With Chronic SCI
Number analyzed (Participants) | 12
g | 0.063 [-0.071 to 0.706]

4. Secondary Outcome: Change in Serum Bone Biomarkers (CTX and P1NP)
Description: Change from baseline to the Month 12 visit in serum levels of CTX and P1NP.
Time Frame: Baseline - 12 months
Population: Females with chronic SCI
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Females With Chronic SCI
Number analyzed (Participants) | 12
ng/mL
  CTX | -0.0093 [-0.048 to 0.025]
  P1NP | -18.25 [-23.56 to -4.27]

ADVERSE EVENTS:
Time Frame: 25 months
Description: Adverse events were obtained by asking participants about changes in their health status during the course of the study. A MedDRA database was used to document all adverse events. Reports of safety outcomes were generated for use by the data and safety monitoring committee (DSMC) to review. DSMC meetings occured at least every 6 months. All serious adverse events (SAEs) were reported as required to the local IRB, Amgen, and FDA.
Groups:
- Year 1: Romosozumab: Participants received monthly subcutaneous injections of romosozumab (210 mg) for 12 months.
- Year 2: Alendronate: Participants received alendronate (70 mg, oral, weekly) for an additional 12 months.
Arm/Group | Year 1: Romosozumab | Year 2: Alendronate
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 2/12
Other Adverse Events (participants affected / at risk) | 12/12 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Year 1: Romosozumab (N=12) | Year 2: Alendronate (N=12)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Year 1: Romosozumab (N=12) | Year 2: Alendronate (N=12)
Injection site reaction (General disorders) | 8 (14) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Urinary tract infection (UTI) (Renal and urinary disorders) | 4 (5) | 2 (3)
Burn (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anisocoria (Eye disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
COVID-19 viral infection (Infections and infestations) | 5 (5) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Spasticity (Nervous system disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1)
Laceration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Upper respiratory infection (cold) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Edema, ankle (General disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Onycholysis of toe (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Thromboembolic event (PE or DVT) (Vascular disorders) | 1 (1) | 0 (0)
Surgical site bleeding (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Left knee injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 2 (2) | 0 (0)
Low phosphorous level (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Peripheral neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 1 (1)
Bilateral ankle abrasions (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Right ankle sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abscess to left buttock (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Right hip subluxation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mild asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Edema, limbs (General disorders) | 0 (0) | 1 (1)
Aortic valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Hemarthrosis of left knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cool right lower extremity (Vascular disorders) | 0 (0) | 1 (1)
Abrasions (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bladder calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Ear infection (otitis media) (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Respiratory syncytial virus (RSV) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne vulgaris of buttock (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Heartburn/Acid Reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fracture of ribs (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT04708886/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT04708886/ICF_001.pdf